CLINICAL TRIAL: NCT00358891
Title: Follow-Up of Very Low Birth Weight Preterm Infants With Chronic Lung Disease at Preschool Ages: Respiratory Health and Neurodevelopment
Brief Title: Follow-Up of VLBW Infants With Chronic Lung Disease: Respiratory Health and Neurodevelopment
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Other Study IDs: 9461701282
Record Dates: First submitted 2006-07-30; First posted 2006-08-01 (Estimated); Last update posted 2006-08-02 (Estimated); Status verified 2006-07

CONDITIONS: Premature Birth
Keywords: Prematurity; Chronic Lung Disease; Respiratory Health; Neurodevelopment; Preschool; Influencing Factors
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Although previous studies showed that preterm infants resolving from neonatal respiratory disease are more likely to exhibit respiratory illness, developmental disorders, impaired growth and cognitive limitations compared with those without, the information concerning the longitudinal respiratory and neurodevelopmental outcome of recently survived preterm infants with CLD is limited.Therefore, the purpose of this study is threefold. First, VLBW infants with CLD, VLBW infants without CLD and full-term infants will be examined for respiratory health at 3-5 years old and will be assessed the relations of early respiratory and environmental variables with later respiratory outcome. Secondly, all infants will be examined for neurodevelopmental outcome, and will be assessed the relations of early neuromotor and environmental variables with later neurodevelopmental outcome. Thirdly, the VLBW infants will be assessed for the concurrent and consecutive longitudinal relationships between respiratory and neurodevelopmental measures.

DETAILED DESCRIPTION:
The introduction of antenatal steroid use, postnatal surfactant administration and modern respiratory care in the past decade has markedly improved the survival of small preterm infants. However, this has been offset by an increasing incidence of chronic lung disease CLD) as defined by oxygen requirement at 36 weeks post-conceptional age. Although previous studies showed that preterm infants resolving from neonatal respiratory disease are more likely to exhibit respiratory illness, developmental disorders, impaired growth and cognitive limitations compared with those without, the information concerning the longitudinal respiratory and neurodevelopmental outcome of recently survived preterm infants with CLD is limited. Therefore, this prospective three-year two-centered study will continue following up the respiratory health and neurodevelopment of our 73 very low birth weight (VLBW) preterm infants at preschool ages. This cohort consists of 44 infants with CLD and 29 demographically matched infants without CLD who were enrolled from the National Taiwan University Hospital and the MacKay Memorial Hospital. Those infants had been comprehensively examined for their respiratory function and neurodevelopmental performance during the neonatal and infant periods. Twenty five age-matched full-term infants will be additional included to serve as the normal reference group. The purpose of this study is threefold. First, VLBW infants with CLD, VLBW infants without CLD and full-term infants will be examined for respiratory health using pulmonary function and exercise test at 3-5 years old and will be assessed the relations of early respiratory and environmental variables with later respiratory outcome. Secondly, all infants will be examined for neurodevelopmental outcome using the Bayley Scales of Infant Development- 2nd edition, Developmental Test of Visual Motor Integration, Peabody Developmental Motor Scale- 2nd edition, Child Behavior Check List, Weschler Preschooler Intelligence Scale and clinical diagnosis by a pediatric neurologist and a pediatric psychiatrist, and will be assessed the relations of early neuromotor and environmental variables with later neurodevelopmental outcome. Thirdly, the VLBW infants will be assessed for the concurrent and consecutive longitudinal relationships between respiratory and neurodevelopmental measures. The results of this study will help understand the nature and changes of respiratory health and neurodevelopment of VLBW infants with CLD from birth to preschool age. The identified influencing factors for adverse respiratory and neurodevelopmental outcome will assist health professionals in designing treatment strategies to improve their outcome. Furthermore, the obtained database will help develop a national monitoring system for measuring effects of respiratory management and early intervention programs for preterm infants with neonatal respiratory disease.

ELIGIBILITY:
Inclusion Criteria:

* BW below 1,500 gm
* GA under 34 weeks
* Admission to the NTUH and MMH within the first 7 days

Exclusion Criteria:

* Existence of congenital anomalies and genetic disease

Ages: 0 Years to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98
Dates: Start 2006-08; Study Completion 2009-07

CONTACTS AND LOCATIONS:
Overall Officials: Suh-Fang Jeng, Sc.D, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Li SJ, Tsao PN, Tu YK, Hsieh WS, Yao NJ, Wu YT, Jeng SF. Cognitive and motor development in preterm children from 6 to 36 months of age: Trajectories, risk factors and predictability. Early Hum Dev. 2022 Sep;172:105634. doi: 10.1016/j.earlhumdev.2022.105634. Epub 2022 Jul 28. PMID 35921693